CLINICAL TRIAL: NCT04527003
Title: A Randomized Controlled Pilot Study of the Use of Cannabidiol in the Management of Endometriosis Pain
Brief Title: Cannabidiol and Management of Endometriosis Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment has been challenging due to the BMI cutoff, need to take oral progesterone and abstain from cannabis products prior to the study.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kristin Riley, MD, Assistant Professor of Obstetrics and Gynecology, Penn State Health Milton S Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00013752
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis; CBD; Pelvic Pain
Keywords: endometriosis; CBD; pelvic pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Cannabidiol; Norethindrone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind of study team (PI, Sub-I's and all research staff) and subjects. Randomization will be completed by Investigational Pharmacy and will keep the blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A - Placebo (Placebo Comparator): Norethindrone acetate (5mg daily) + Placebo
  Interventions: Drug: Norethindrone Acetate; Other: Placebo
- Group B - Low Dose CBD (Active Comparator): Norethindrone acetate (5mg daily) + Low dose CBD (10mg sublingual daily)
  Interventions: Drug: Cannabidiol (CBD) Extract; Drug: Norethindrone Acetate
- Group C - High Dose CBD (Active Comparator): Norethindrone acetate (5mg daily) + High dose CBD (20mg sublingual daily)
  Interventions: Drug: Cannabidiol (CBD) Extract; Drug: Norethindrone Acetate

INTERVENTIONS:
Drug: Cannabidiol (CBD) Extract — Cannabis is a well-known plant that contains more than 500 identified phytochemicals of which over 100 are cannabinoids. The most widely studied is 9-tetrahydrocannabinol (9-THC), which is the major psychoactive component of Cannabis, but Cannabidiol (CBD) has been increasingly favored for its reduced side effect profile and potential health benefits. CBD was first isolated from Cannabis in the 1940s. CBD, unlike 9-THC, does not bind to CB1 and CB2 receptors, which accounts for its lack of typical psychotropic effects, but is still appears to work via alternative mechanisms via the endocannabinoid system.
  Arms: Group B - Low Dose CBD; Group C - High Dose CBD
Drug: Norethindrone Acetate — Norethindrone is a form of progesterone, a female hormone important for regulating ovulation and menstruation.
Other: Placebo — a substance or treatment which is designed to have no therapeutic value
  Arms: Group A - Placebo

SUMMARY:
The investigators are looking to conduct a study looking at the effects of cannabidiol (CBD) in patients with endometriosis. It is believed that CBD will improve both pain and quality of life. The study will last a total of 12 weeks and involve several onsite visits in addition to daily pain assessments.

DETAILED DESCRIPTION:
The proposal is to conduct a randomized double-blind placebo-controlled pilot study to evaluate the effectiveness of cannabidiol on the management of endometriosis-related pain.

Subjects will be pre-screened from new and existing patients as well as from referral sites for the diagnosis of endometriosis. Potential subjects will be pre-screened for moderate to severe endometriosis associated pain (VAS > 3) greater than 6 months. Those meeting all inclusion and exclusion criteria that who are willing to participate will receive a detailed history and physical exam, appropriate bloodwork and undergo informed consented at the Screening Visit. Baseline survey data will be collected. During Screening, the patient's will be asked to complete their daily electronic diaries and screened for daily reporting adherence.

Randomized subjects will receive either (1) placebo (2) low dose CBD (3) high dose CBD. This study will include an 8-week intervention period during which subjects will be asked to record daily electronic VAS scores, pain medication use and a number of other parameters. Subjects will return at week 12 for a 4 week post-treatment visit, where they can also chose to enroll in an optional pharmacokinetic study. Participants will complete the Endometriosis Health Profile-30 (EHP-30), Patient Global Assessments (PGAs), the Patient Global Impression of Change (PGIC) surveys and, if partnered and sexually active, the Female Sexual Function Index at various time points. Patients will also have bloodwork done to assess for circulating markers of inflammation, circulating CBD concentration levels and liver dysfunction throughout the study duration. Subjects will be screened for side effects and asked to record pain medication use throughout the duration of the study. Study drug compliance will be assessed.

At the completion of the study, all subjects will be offered the opportunity to do pharmacokinetic testing with sublingual CBD until a maximum number of 4 patients are enrolled. The testing will include 24 hours of monitoring with sequential blood draws to determine the pharmacokinetic parameters of sublingual CBD after administration and one salivary pH. They will be discharged at 24 hours and asked to return to the clinic at 48 hours for one final lab draw.

ELIGIBILITY:
Inclusion Criteria:

1. Females ages 18-45 years at the time of enrollment
2. A surgical diagnosis with direct visualization and/or histopathologic confirmation of endometriosis with associated moderate to severe endometriosis related pain ( > 3 on a VAS)
3. Is not expected to undergo gynecological surgery or other surgical procedure for treatment of endometriosis during the study period
4. Agrees to use approved contraception during the entire study if not surgically sterile
5. Patients using oral contraceptives, vaginal ring, injectable progesterone and/or GnRH agonists/antagonist for contraception and/or management of endometriosis, can be included if both they and their primary provider agree to stopping their medication and transitioning to Norethindrone acetate (NETA) as the primary treatment of endometriosis throughout the study period.
6. Patients using Long-acting reversible contraceptives (LARCs) for contraception and/or management of endometriosis can be included if both they and their primary provider agree to initiate Norethindrone (NETA) as the primary treatment of endometriosis throughout the study period

Exclusion Criteria:

1. Women that are pregnant, breastfeeding or trying to conceive
2. Women with chronic daily opioid use and any chronic pain or frequently reoccurring pain condition, other than endometriosis, that is treated with opioids for > 14 days per month.
3. Women that are currently using Cannabis based products or have used them within 30 days of enrollment
4. Non-English speaking or inability to read and understand English
5. Women with a BMI > 35 kg/m2
6. Women with known liver disease, such as hepatitis, or with screening LFTS (AST/ALT) > 3 times above the upper limits of normal (ULN) in the past year
7. Women with chronic alcohol use (defined as > 3 drinks per day, averaged over one week)
8. Women with chronic use of drugs (defined as > 10 days/month) that cause somnolence/sedation such as benzodiazepines or Central Nervous System (CNS) depressants that are unwilling or unable to discontinue the medications for the washout period and the duration of the study
9. Women who are currently taking Clobazam or Valproate and are unwilling/unable to discontinue the medication for the washout period and the duration of the study
10. Women with suicidal ideation or uncontrolled depression within the past year
11. Known history of or suspected breast cancer on screening physical exam
12. History of or active deep venous thrombosis or pulmonary embolism
13. History of or active arterial thromboembolic event (e.g. stroke, myocardial infarction)
14. Multiple (> 3) risk factors for arterial vascular disease (e.g. uncontrolled hypertension, diabetes mellitus, hypercholesterolemia, obesity and smoking)
15. Current use of a progestin-containing contraceptive implant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females ages 18-45 years at the time of enrollment who have a surgical diagnosis with direct visualization and/or histopathologic confirmation of endometriosis with associated moderate to severe endometriosis related pain
Enrollment: 12 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burney RO, Giudice LC. Pathogenesis and pathophysiology of endometriosis. Fertil Steril. 2012 Sep;98(3):511-9. doi: 10.1016/j.fertnstert.2012.06.029. Epub 2012 Jul 20. PMID 22819144
- [Background] Giudice LC, Kao LC. Endometriosis. Lancet. 2004 Nov 13-19;364(9447):1789-99. doi: 10.1016/S0140-6736(04)17403-5. PMID 15541453
- [Background] Behera M, Vilos GA, Hollett-Caines J, Abu-Rafea B, Ahmad R. Laparoscopic findings, histopathologic evaluation, and clinical outcomes in women with chronic pelvic pain after hysterectomy and bilateral salpingo-oophorectomy. J Minim Invasive Gynecol. 2006 Sep-Oct;13(5):431-5. doi: 10.1016/j.jmig.2006.05.007. PMID 16962527
- [Background] Rafique S, Decherney AH. Medical Management of Endometriosis. Clin Obstet Gynecol. 2017 Sep;60(3):485-496. doi: 10.1097/GRF.0000000000000292. PMID 28590310
- [Background] Lamvu G, Soliman AM, Manthena SR, Gordon K, Knight J, Taylor HS. Patterns of Prescription Opioid Use in Women With Endometriosis: Evaluating Prolonged Use, Daily Dose, and Concomitant Use With Benzodiazepines. Obstet Gynecol. 2019 Jun;133(6):1120-1130. doi: 10.1097/AOG.0000000000003267. PMID 31135725
- [Background] Fasinu PS, Phillips S, ElSohly MA, Walker LA. Current Status and Prospects for Cannabidiol Preparations as New Therapeutic Agents. Pharmacotherapy. 2016 Jul;36(7):781-96. doi: 10.1002/phar.1780. PMID 27285147
- [Background] Hermanson DJ, Marnett LJ. Cannabinoids, endocannabinoids, and cancer. Cancer Metastasis Rev. 2011 Dec;30(3-4):599-612. doi: 10.1007/s10555-011-9318-8. PMID 22038019
- [Background] Bouaziz J, Bar On A, Seidman DS, Soriano D. The Clinical Significance of Endocannabinoids in Endometriosis Pain Management. Cannabis Cannabinoid Res. 2017 Apr 1;2(1):72-80. doi: 10.1089/can.2016.0035. eCollection 2017. PMID 28861506
- [Background] Brawn J, Morotti M, Zondervan KT, Becker CM, Vincent K. Central changes associated with chronic pelvic pain and endometriosis. Hum Reprod Update. 2014 Sep-Oct;20(5):737-47. doi: 10.1093/humupd/dmu025. Epub 2014 Jun 11. PMID 24920437
- [Background] Rocha MG, e Silva JC, Ribeiro da Silva A, Candido Dos Reis FJ, Nogueira AA, Poli-Neto OB. TRPV1 expression on peritoneal endometriosis foci is associated with chronic pelvic pain. Reprod Sci. 2011 Jun;18(6):511-5. doi: 10.1177/1933719110391279. Epub 2010 Dec 15. PMID 21160085
- [Background] Bohonyi N, Pohoczky K, Szalontai B, Perkecz A, Kovacs K, Kajtar B, Orban L, Varga T, Szegedi S, Bodis J, Helyes Z, Koppan M. Local upregulation of transient receptor potential ankyrin 1 and transient receptor potential vanilloid 1 ion channels in rectosigmoid deep infiltrating endometriosis. Mol Pain. 2017 Jan-Dec;13:1744806917705564. doi: 10.1177/1744806917705564. PMID 28478727
- [Background] Sanchez AM, Vigano P, Mugione A, Panina-Bordignon P, Candiani M. The molecular connections between the cannabinoid system and endometriosis. Mol Hum Reprod. 2012 Dec;18(12):563-71. doi: 10.1093/molehr/gas037. Epub 2012 Aug 24. PMID 22923487
- [Background] Devinsky O, Verducci C, Thiele EA, Laux LC, Patel AD, Filloux F, Szaflarski JP, Wilfong A, Clark GD, Park YD, Seltzer LE, Bebin EM, Flamini R, Wechsler RT, Friedman D. Open-label use of highly purified CBD (Epidiolex(R)) in patients with CDKL5 deficiency disorder and Aicardi, Dup15q, and Doose syndromes. Epilepsy Behav. 2018 Sep;86:131-137. doi: 10.1016/j.yebeh.2018.05.013. Epub 2018 Jul 11. PMID 30006259
- [Background] Ewing LE, Skinner CM, Quick CM, Kennon-McGill S, McGill MR, Walker LA, ElSohly MA, Gurley BJ, Koturbash I. Hepatotoxicity of a Cannabidiol-Rich Cannabis Extract in the Mouse Model. Molecules. 2019 Apr 30;24(9):1694. doi: 10.3390/molecules24091694. PMID 31052254
- [Background] Millar SA, Stone NL, Yates AS, O'Sullivan SE. A Systematic Review on the Pharmacokinetics of Cannabidiol in Humans. Front Pharmacol. 2018 Nov 26;9:1365. doi: 10.3389/fphar.2018.01365. eCollection 2018. PMID 30534073
- [Background] Lucas CJ, Galettis P, Schneider J. The pharmacokinetics and the pharmacodynamics of cannabinoids. Br J Clin Pharmacol. 2018 Nov;84(11):2477-2482. doi: 10.1111/bcp.13710. Epub 2018 Aug 7. PMID 30001569
- [Background] Roslawski MJ, Remmel RP, Karanam A, Leppik IE, Marino SE, Birnbaum AK. Simultaneous Quantification of 13 Cannabinoids and Metabolites in Human Plasma by Liquid Chromatography Tandem Mass Spectrometry in Adult Epilepsy Patients. Ther Drug Monit. 2019 Jun;41(3):357-370. doi: 10.1097/FTD.0000000000000583. PMID 30520828
- See also: HIGHLIGHTS OF PRESCRIBING INFORMATION. EPIDIOLEX ® (cannabidi ol) oral solution, CX [pending DEA scheduling action] Initial U.S. Approval: XXXX [pending controlled substance scheduling] — http://www.fda.gov

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between screening and randomization, subjects entered a run-in phase collecting daily electronic diaries. Subjects were excluded from randomization if they were not at least 80% adherent with completion of the daily diaries.
Period: Overall Study
Arm/Group | Group A - Placebo | Group B - Low Dose CBD | Group C - High Dose CBD
Started | 4 | 3 | 3
Completed | 4 | 2 | 1
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Placebo | Group B - Low Dose CBD | Group C - High Dose CBD | Total
Number analyzed (Participants) | 4 | 3 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (6.2) | 24.4 (7.3) | 28.9 (5.4) | 28.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 3 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Area Under the Curve (AUC)
Description: Pain will be self-reported daily using the Visual Analog Scale, a 100mm horizontal line on which the patient's pain intensity is represented by a point between the extremities of 0 (no pain) and 100 (worst pain). Although the daily collection is based on the 0-100 point scale, the primary study endpoint is calculated as the area under the curve per patient using the trapezoidal rule, with an AUC range per patient of 0-5600 over 8 weeks.
Time Frame: 8 weeks
Population: Subjects who completed the study
Measure: Median (Inter-Quartile Range); unit: score on a scale*days
Arm/Group | Group A - Placebo | Group B - Low Dose CBD | Group C - High Dose CBD
Number analyzed (Participants) | 4 | 2 | 1
score on a scale*days | 2254 [1803 to 2662] | 2211 [1455 to 2968] | 1042 [1042 to 1042]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: At follow-up visits (4 weeks, 8 weeks, 12 weeks), adverse event assessment will include, but is not limited to:
  1. Detailed, directed review of systems
  2. Vital signs
  3. Examination of oral cavity (to assess for lesions/sores)
  4. Physical exam
Arm/Group | Group A - Placebo | Group B - Low Dose CBD | Group C - High Dose CBD
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Placebo (N=4) | Group B - Low Dose CBD (N=3) | Group C - High Dose CBD (N=3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headaches (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Gagging (when taking study drug) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
ulcer on lip (General disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study struggled with recruitment and terminated early, leading to very small numbers of subjects per treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT04527003/Prot_SAP_000.pdf